CLINICAL TRIAL: NCT03903029
Title: AssessmeNt of Efficacy of Low-dose rosuvaStatin in KoRean 4 Statin Benefit Groups Per 2013 ACC/AHA Guideline
Brief Title: Efficacy of Low-dose (10 mg) Rosuvastatin in Korean 4 Statin Benefit Groups Per 2013 ACC/AHA Guideline
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NewStaR4G
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Dyslipidemias
Keywords: Cholesterol, LDL; Asian; Rosuvastatin; Low-dose
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low-dose (10mg) rosuvastatin: Four statin benefit groups per 2013 ACC/AHA guideline in Korea
  Interventions: Drug: Low-dose (10mg) rosuvastatin

INTERVENTIONS:
Drug: Low-dose (10mg) rosuvastatin — Low-dose (10mg) rosuvastatin in 4 statin benefit groups per 2013 ACC/AHA guideline
  Other Names: Crestor

SUMMARY:
This study aimed to evaluate the efficacy of low-dose rosuvastatin (10 mg) in the 4 statin benefit groups requiring high- or moderate-intensity statin therapy according to the 2013 American College of Cardiology/American Heart Association guideline in Korean population.

DETAILED DESCRIPTION:
The primary endpoint was percentage reduction in low-density lipoprotein (LDL) cholesterol. Secondary endpoints were percentage reduction in other lipids and achievement of ≥50% reduction in LDL cholesterol. Intention-to-treat analyses were performed.

ELIGIBILITY:
Inclusion Criteria:

1. subjects with prior history of clinical ASCVD
2. subjects with primary elevation of LDL cholesterol ≥190 mg/dL
3. subjects with diabetes, age 40 to 75 years, and LDL cholesterol 70 to 189 mg/dL
4. subjects without diabetes, age 40 to 75 years, LDL cholesterol 70 to 189 mg/dL, and with estimated 10-year ASCVD risk ≥7.5%.

Exclusion Criteria:

1. history of significant statin-induced rhabdomyolysis or myopathy
2. history of a significant hypersensitivity reaction to rosuvastatin
3. uncontrolled diabetes mellitus (HbA1c >9%)
4. uncontrolled hypertension (systolic blood pressure >190 mmHg or diastolic blood pressure >100 mmHg)
5. current active liver disease (alanine aminotransferase and/or aspartate aminotransferase >2 times the upper limit of normal)
6. chronic kidney disease (serum creatinine clearance <30 ml/min)
7. creatine kinase levels >3 times the upper limit of normal
8. use of prohibited concomitant therapies
9. history of malignancy within the last 5 years
10. women who were pregnant, breast-feeding or of childbearing potential without contraception
11. subjects who would take any medication for purposes other than this trial within 30 days after taking this study's medication.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four statin benefit groups per 2013 ACC/AHA guideline in Korean
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2015-07-05 (Actual); Study Completion 2019-12-05 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction in low-density lipoprotein (LDL) cholesterol | 8 weeks
  Percentage reduction in low-density lipoprotein (LDL) cholesterol from baseline to 8 weeks of treatment

SECONDARY OUTCOMES:
Percentage reduction in other lipids | 8 weeks
  Percent changes from baseline to 8 weeks in total cholesterol, high-density lipoprotein (HDL) cholesterol, triglyceride (TG), non-HDL cholesterol, apolipoprotein B, apolipoprotein A1
Achievement of ≥50% reduction in LDL cholesterol | 8 weeks
  Achievement of ≥50% reduction in LDL cholesterol with use of rosuvastatin 10 mg in 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD., PhD., Study Chair — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No